CLINICAL TRIAL: NCT00303199
Title: A Phase I/II Trial of ZIO-101 in Advanced Multiple Myeloma
Brief Title: Study of ZIO-101 in Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGL2001
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Arsenic; Cancer study; Failed treatment
MeSH Terms: conditions — Multiple Myeloma | interventions — darinaparsin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: ZIO-101 (Darinaparsin)

INTERVENTIONS:
Drug: ZIO-101 (Darinaparsin) — IV zio-101 (Darinaparsin) give for 5 consecutive days to be repeated every 28 days for up to 6 months
  Other Names: ZIO-101

SUMMARY:
The study of safety of a new organic arsenic compound in the treatment of advanced multiple myeloma

ELIGIBILITY:
Subjects with multiple myeloma who have received at least two prior therapies and currently require therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Phase I: toxicity defined in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v3.0 (CTCAE) 12/12/03 | 6 months
Phase II efficacy using EMBT criteria. | 6 months
Safety | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics of ZIO-101 | 6 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Little Rock, Arkansas
  - West Hollywood, California
  - Miami, Florida
  - Bethesda, Maryland
  - New York, New York
  - Cleveland, Ohio
- Canada (2):
  - Edmonton, Alberta
  - Toronto, Ontario